CLINICAL TRIAL: NCT04155047
Title: A Randomized, Double-blind, Placebo-controlled, 2-Way Crossover Study of the Effect of a Single Dose of Glycopyrrolate Inhalation Solution (GIS) on Lung Hyperinflation in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Clinical Study to Investigate if a Single Dose of an Approved Drug Product (Glycopyrrolate Inhalation Solution) Reduces Trapped Air in the Lungs of Participants With Chronic Obstructive Pulmonary Disease.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunovion Respiratory Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: SUN101-402
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-blind, Placebo-controlled, 2-Way Crossover Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Glycopyrrolate Inhalation Solution (Active Comparator): Glycopyrrolate Inhalation Solution 25mcg administered by Magnair
  Interventions: Combination Product: Glyocopyrrolate Inhalation Solution administered by Magnair
- Placebo (Placebo Comparator): Placebo Inhalation Solution administered by Magair
  Interventions: Drug: Placebo administered by Magnair

INTERVENTIONS:
Combination Product: Glyocopyrrolate Inhalation Solution administered by Magnair — glycopyrrolate Inhalation Solution 25mcg, single dose
  Other Names: LONHALA
  Arms: Glycopyrrolate Inhalation Solution
Drug: Placebo administered by Magnair — Placebo Inhalation Solution
  Arms: Placebo

SUMMARY:
A clinical study to investigate if a single dose of an approved drug product (glycopyrrolate Inhalation Solution) reduces trapped air in the lungs of participants with chronic obstructive pulmonary disease. This study is accepting male and female participants over the age of 40. The study will be conducted at one site located in the United States.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, placebo-controlled, single-dose, 2-way crossover study in approximately 20 adult subjects ≥ 40 years of age with COPD. The study is designed to evaluate the effect of a single dose of GIS on lung hyperinflation. The two study treatments, both administered using the Magnair device.

The study will randomize 10 subjects per treatment sequence, for a total of 20 subjects. At the Sponsor's discretion, additional subjects may be enrolled in an effort to achieve at least 20 completers, with no more than 24 subjects randomize.

The study will consist of a Screening period, a randomized 2-way cross-over treatment period during which subjects will receive two single-doses each separated by a 7-day washout period, and a follow-up 7 (± 2) days after the last study drug dose.

This study is designed to test the hypothesis that in adults with COPD subjects as characterized by the study inclusion/exclusion criteria, after 2 cross-over periods of treatment, the primary null hypothesis for this study is that the mean change of RV from baseline at 6 hours postdose for a single dose of GIS is equal to the mean change of RV from baseline at 6 hours postdose for a single dose of placebo inhalation solution (PIS). The alternative hypothesis is that these means are different.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female and ≥ 40 years of age at Screening with a confirmed diagnosis of COPD.

Subject must have the ability to comprehend the informed consent form and be willing to provide informed consent.

Subject must possess an educational level and degree of understanding of English that enables them to communicate suitably with the Investigator and the study coordinator.

Subject has a postbronchodilator (following inhalation of ipratropium bromide) FEV1 ≥ 30% and < 80% of predicted normal at Screening.

Subject has a postbronchodilator (following inhalation of ipratropium bromide) FEV1/FVC ratio of < 0.70 at Screening.

Subject has a RV ≥ 130% predicted value at Screening (prior to reversibility testing) Subject is a current or former smoker with at least 10 pack-years of cigarette smoking history at Screening.

Subject has a score of ≥ 2 on the Modified Medical Research Council Dyspnea Scale (mMRC) at Screening.

Subject, if female of child bearing potential, must have a negative serum pregnancy test at Screening. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control: a) an oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 30 days prior to entering the study with continued use throughout the study and for thirty days following participation; b) barrier method of contraception, eg, condom and /or diaphragm with spermicide while participating in the study; and/or c) abstinence. A follicle stimulating hormone (FSH) test will be used to confirm menopause in postmenopausal females.

Subject is willing and able to attend all study visits and adhere to all study assessments and procedures.

* Exclusion Criteria:

Subject is female who is pregnant or lactating or are planning on becoming pregnant during the study.

Subject has a history of asthma. Subject has a blood eosinophil count > 5% of total white blood cell count. Subject has life-threatening/unstable respiratory status, including upper or lower respiratory tract infection, within the previous 30 days prior to Screening.

Recent history of COPD exacerbation requiring hospitalization or need for increased treatments for COPD within 12 weeks prior to Screening.

Use of daily oxygen therapy > 12 hours per day Subject is unable to perform plethysmography. Subject is unable to use the Magnair Nebulizer System. Subject has history of narrow angle glaucoma Subject has history of or clinically significant ongoing bladder outflow obstruction or history of catheterization for relief of bladder outflow obstruction within the previous 6 months prior to screening.

subject has history of long QT syndrome. subject has a QTcF > 450 msec (males) or > 470 msec (females) at Screening, unless discussed with and approved by the Medical Monitor.

Subject has a cardiac implanted device (internal defibrillator, pacemaker). Current severe heart failure (New York Heart Association Class IV) [New York Heart Association, 1994].

Subject has history of malignancies within the past 5 years, with the exception of basal cell carcinoma.

Subject has known comorbidities including unstable cardiac, pulmonary, or psychiatric disease, or any other medical conditions that would, in the opinion of the Investigator, preclude the subject from safely completing the required tests or the study, or is likely to result in disease progression that would require withdrawal of the subject.

Subject has participated in another investigational drug study (within 30 days prior to Screening).

Subjects who are study site staff members or relatives of study site staff members.

Subjects with a history of allergic reaction to glycopyrrolate, tiotropium, albuterol, or any components of the study medications.

Subjects with a known allergy to hydrocolloid gel adhesive are excluded from wearing the VitalPatch Biosensor.

-Continuation Criteria Subject has not had an exacerbation of COPD. Subject completes the 7-day washout period and continues to withhold restricted medications.

In the opinion of the Investigator, the subject has not had any change that would put the safety of the subject at risk through participation.

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Respiratory Medical Director, Study Chair — Sumitomo Pharma America, Inc.
Locations (1):
- Midwest Chest Consultants, Saint Charles, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study may be made available upon request via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available upon request within 12 months of posting the study results on ct.gov.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Siler TM, Hohenwarter C, Xiong K, Sciarappa K, Sanjar S, Sharma S. Efficacy of Nebulized Glycopyrrolate on Lung Hyperinflation in Patients with COPD. Pulm Ther. 2021 Dec;7(2):503-516. doi: 10.1007/s41030-021-00166-5. Epub 2021 Jul 7. PMID 34232493

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 44 subjects enrolled in the study. There were 22 subjects that screen failed and did not participate in the study. There were 22 subjects that started the study.
Groups:
- Glycopyrrolate Inhalation Solution (GIS) First, Then Placebo Inhalation Solution (PIS): Treatment sequence AB: Single dose of GIS 25 mcg (Treatment A) to matching PIS (Treatment B)
- Placebo Inhalation Solution (PIS) First, Then Glycopyrrolate Inhalation Solution (GIS): Treatment sequence BA: Matching PIS (Treatment B) to single dose of GIS 25 mcg (Treatment A)
Period: Overall Study
Arm/Group | Glycopyrrolate Inhalation Solution (GIS) First, Then Placebo Inhalation Solution (PIS) | Placebo Inhalation Solution (PIS) First, Then Glycopyrrolate Inhalation Solution (GIS)
Started | 11 | 11
Completed | 9 | 11
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — COVID-19: SUBJECT REFUSED STUDY VISITS DUE TO COVID-19 THREAT | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glycopyrrolate Inhalation Solution (GIS) First, Then Placebo Inhalation Solution (PIS) | Placebo Inhalation Solution (PIS) First, Then Glycopyrrolate Inhalation Solution (GIS) | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.4 (8.03) | 66.5 (8.12) | 65.9 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight (kg) [Mean (Standard Deviation); unit: kg] | 96.69 (22.683) | 92.65 (23.808) | 94.67 (22.785)
Height (cm) [Mean (Standard Deviation); unit: cm] | 166.4 (12.18) | 175.1 (8.94) | 170.8 (11.33)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 34.67 (6.131) | 30.14 (7.086) | 32.4 (6.87)
Baseline Residual Volume for GIS 25 mcg [Mean (Standard Deviation); unit: L] | 3.132 (0.5631) | 3.696 (0.7570) | 3.414 (0.7123)
Baseline Residual Volume for Placebo [Mean (Standard Deviation); unit: L] — Population: Among the 11 participants in treatment sequence AB, 2 participants received Treatment A (GIS 25mcg) in period 1 and did not continue into period 2. Therefore, there were only 9 participants with baseline measures for Treatment B (PIS).
  L
    number analyzed (Participants) | 9 | 11 | 20
    (all) | 3.174 (0.5669) | 3.592 (0.6915) | 3.404 (0.6575)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Residual Volume (RV) at 6 Hours Postdose
Description: Change from baseline in Residual Volume (Residual Volume is defined as the volume of gas that remains in lungs after maximal exhalation) at 6 hours postdose.
Time Frame: 6 hours post dose
Population: Efficacy Population : all subjects who were randomized, received at least one dose of study treatment, and have a baseline and at least one post-baseline RV measurement within the same period.
Measure: Least Squares Mean (Standard Error); unit: L
Groups:
- Placebo: Placebo Inhalation Solution (PIS) administered by Magair
- GIS 25 mcg Single Dose: Glycopyrrolate Inhalation Solution (GIS) 25 mcg administered by Magnair
Arm/Group | Placebo | GIS 25 mcg Single Dose
Number analyzed (Participants) | 20 | 22
L | 0.004 (0.1392) | -0.319 (0.1313)
Statistical Analysis 1: Comparison: Placebo vs GIS 25 mcg Single Dose; Test type: Superiority; p = 0.0987, Mixed Models Analysis; Least Squares Mean Difference = -0.323, 95% CI 2-sided [-0.711 to 0.066], Standard Error of Mean 0.1861

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Placebo | GIS 25 mcg Single Dose
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 0/20 | 1/22
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | GIS 25 mcg Single Dose (N=22)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT04155047/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT04155047/SAP_001.pdf